CLINICAL TRIAL: NCT00643279
Title: Chronicle Offers Management to Patients With Advanced Signs and Symptoms of Heart Failure (COMPASS-HF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: COMPASS-HF
Record Dates: First submitted 2008-02-29; First posted 2008-03-26 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure
Keywords: implantable hemodynamic monitor; Intracardiac pressures
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHRONICLE (Experimental): Subjects randomized to the CHRONICLE group were managed using data from an implantable hemodynamic monitoring (IHM) device, including trended right ventricular (RV) and estimated pulmonary arterial (PA) pressures, heart rate and activity data. The Chronicle IHM device does not provide therapy, but rather provides intracardiac diagnostic information about the patient which the physician can utilize to manage the patient and the patients heart failure.
  Interventions: Device: Chronicle Implantable Hemodynamic Monitor
- CONTROL (Placebo Comparator): Subjects randomized to the CONTROL group implanted with the Chronicle implantable hemodynamic monitoring (IHM) device, but the intracardiac diagnostic information was blinded to both the patient and the physician during the randomized period of the study. Subjects were managed conventionally with standard of care. Physicians and patients have access to the intracardiac data after the randomized period of the study is over, at 6 months.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Chronicle Implantable Hemodynamic Monitor — Surgical implantation of chronic ambulatory implantable hemodynamic monitoring (IHM) device and intracardiac pressure sensing lead. The implantable hemodynamic monitoring device captures intracardiac hemodynamic information about the patient including trended right ventricular (RV) and estimated pulmonary arterial (PA) pressures, heart rate and activity data. The IHM device does not provide therapy, but rather provides intracardiac diagnostic information about the patient which the physician can utilize to manage the patient and the patients heart failure.
  Arms: CHRONICLE
Other: Standard of Care — Surgical implantation of chronic ambulatory implantable hemodynamic monitoring (IHM) device and intracardiac pressure sensing lead, but physician and patient access to the intracardiac information provided by the device is restricted until the end of the randomized period of the study, at 6 months. Patients and patients heart failure are managed conventionally per standard of care.
  Arms: CONTROL

SUMMARY:
COMPASS-HF was a prospective, two-arm, randomized (1:1), multi-center, parallel controlled study. The purpose of the randomized study was to test the safety of an implantable hemodynamic monitor (IHM) and pressure sensor lead. The premise of this study was to compare the effectiveness of a novel heart failure management strategy based on information obtained from the IHM system in reducing heart failure morbidity compared to a strategy based on standard medical care alone.

DETAILED DESCRIPTION:
COMPASS-HF was a prospective, two-arm, randomized (1:1), multi-center, parallel controlled study. The purpose of the randomized study was to test the safety of an implantable hemodynamic monitor (IHM) and pressure sensor lead. The premise of this study was to compare the effectiveness of a novel heart failure management strategy based on information obtained from the IHM system in reducing heart failure morbidity compared to a strategy based on standard medical care alone.

After baseline evaluation and verification that entrance criteria were met, all subjects were implanted with a Chronicle IHM and pressure sensor lead. Following successful implantation, subjects were randomized to either the CHRONICLE group or CONTROL group. Subjects randomized to the CHRONICLE group were managed using Chronicle, specifically trended RV and estimated PA pressure, heart rate and activity data, whereas subjects randomized to the CONTROL group were treated conventionally without the use of the Chronicle data. In the case that implantation was not successful, subjects were exited from the study if no procedure related adverse events were identified; procedure related adverse events were followed through to resolution before the subject were withdrawn from the study.

Subjects remained randomized until their six month clinic visit had been completed. Following the subject's six month visit, clinicians were granted access to the CONTROL subject's trended Chronicle data on the Chronicle website, and subjects were seen in the clinic for a protocol-required visit every six months until exit from the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with heart failure classified as New York Heart Association (NYHA) Class III and IV
* Subject has been managed with standard medical therapy for heart failure (such as diuretic, angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blockers (ARB), and beta-blocker for at least 3 months prior to the baseline evaluation
* Subject must have at least one heart failure-related hospitalization or emergency department visit requiring intravenous treatment within 6 months prior to baseline evaluation

Exclusion Criteria:

* Subjects who are likely to be transplanted within 6 months from randomization or will remain hospitalized until transplantation
* Subjects with severe COPD or restrictive airway disease (recommended FEV1 less than or equal to 1 liter or 50% predicted)
* Subjects who are on continuous positive inotropic therapy
* Subjects with known atrial or ventricular septal defects
* Subjects with mechanical right heart valves
* Subjects with stenotic tricuspid or pulmonary valves
* Subjects with a presently implanted non-compatible pacemaker or ICD
* Subjects with cardiac resynchronization therapy which has not achieved optimal programming for more than 3 months
* Subjects with a major cardiovascular event within 3 months prior to baseline evaluation
* Subjects with a severe non-cardiac condition limiting 6 month survival
* Subjects with a primary diagnosis of pulmonary artery hypertension
* Subjects with serum creatinine greater than or equal to 3.5 mg/dL or on chronic renal dialysis
* Subjects enrolled in concurrent studies that may confound the results of this study
* Women who are pregnant or with child bearing potential and who are not on a reliable form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2003-03; Primary Completion 2005-06 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bourge, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (28):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Loma Linda University Medical Center, Loma Linda, California
  - UCLA Medical Center, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - University of Florida - Shands, Gainesville, Florida
  - Crawford LongHospital, Atlanta, Georgia
  - Prairie Heart Institute, Springfield, Illinois
  - Parkview Memorial Hospital, Fort Wayne, Indiana
  - New England Medical Center, Boston, Massachusetts
  - St. Paul Heart, Saint Paul, Minnesota
  - Mid America Heart Institute, Kansas City, Missouri
  - Robert Wood Johnson Medical Center, New Brunswick, New Jersey
  - Newark Beth Israel, Newark, New Jersey
  - New York Presbyterian - Columbia, New York, New York
  - Duke University, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oklahoma Cardiovascular Associates, Oklahoma City, Oklahoma
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baptist Memorial Hospital, Germantown, Tennessee
  - St. Thomas Hospital, Nashville, Tennessee
  - St. Luke's Episcopal Hospital/Texas Heart, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Zile MR, Adamson PB, Cho YK, Bennett TD, Bourge RC, Aaron MF, Aranda JM Jr, Abraham WT, Stevenson LW, Kueffer FJ. Hemodynamic factors associated with acute decompensated heart failure: part 1--insights into pathophysiology. J Card Fail. 2011 Apr;17(4):282-91. doi: 10.1016/j.cardfail.2011.01.010. Epub 2011 Feb 26. PMID 21440865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on March 13, 2003 and ended on November 16, 2004. All subjects were exited from the study on April 8, 2013. Twenty-nine US clinical centers participated in the COMPASS-HF study.
Pre-assignment Details: Subjects were required to have a successful implant of the Chronicle® device prior to randomization. 277 subjects had an attempted implant, with 274 successfully implanted and randomized. 3 subjects had unsuccessful implant attempts and were exited prior to randomization.
Groups:
- Treatment: Physicians have access to device-based hemodynamic monitor information to guide patient management
- Control: Physicians do not have access to device-based hemodynamic monitor information to guide patient management
Period: Overall Study
Arm/Group | Treatment | Control
Started | 134 | 140
Completed | 118 | 127
Not Completed | 16 | 13
Not completed — Death | 13 | 11
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 134 | 140 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (14) | 58 (13) | 58 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 50 | 109
  Male | 75 | 90 | 165
Region of Enrollment [Number; unit: participants]
  United States | 134 | 140 | 274
New York Heart Association Class III (NYHA III) [Count of Participants; unit: Participants] | 112 | 122 | 234
New York Heart Association Class IV (NYHA IV) [Count of Participants; unit: Participants] | 22 | 18 | 40

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by the Percentage of Participants Free From System Related Complications Through 6 Months.
Description: A Chronicle IHM system-related complication was defined as any system-related adverse event that occurred during the clinical investigation which is (1) treated with invasive means (including intravenous drug therapy), (2) results in death, (3) results in the explant of any Chronicle IHM component, and/or (4) causes permanent loss of significant function of the implanted system.
  Safety is defined as ≥ 80% of participants experiencing freedom from device related complications through 6 months.
Time Frame: Within 6 months post-implant
Population: The analysis population for safety includes all subjects with an attempted implant of the Chronicle implantable hemodynamic monitoring device, including both successful implanted participants (274) and unsuccessful implanted participants (3). In total 277 participants were assessed for the safety objective.
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects With Attempted Implant: All subjects with an attempted implant of a Chronicle IHM.
Arm/Group | All Subjects With Attempted Implant
Number analyzed (Participants) | 277
Participants | 277
Statistical Analysis 1: Comparison: All Subjects With Attempted Implant; Test type: Superiority — Survival estimate at 6-months; 6-month survival rate = 91.5, 95% CI 1-sided [lower limit 88.7]

2. Primary Outcome: Safety as Measured by the Percentage of Participants Free From Implantable Hemodynamic Monitor Pressure Related Sensor Lead Failures Through 6 Months.
Description: A pressure sensor failure was defined as a recognizable, abrupt, non-physiologic shift in pressure parameters.
  Safety is defined as ≥ 90% of participants free from pressure sensor lead failure through 6 months.
Time Frame: Within 6 months post-implant
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects Successfully Implanted: All subjects successfully implanted with a Chronicle IHM system
Arm/Group | All Subjects Successfully Implanted
Number analyzed (Participants) | 274
Participants | 274
Statistical Analysis 1: Comparison: All Subjects Successfully Implanted; Test type: Superiority — Survival estimate at 6-months; 6-month survival rate = 100, 95% CI 1-sided [lower limit 98.9]

3. Primary Outcome: Rate of Heart Failure-related Hospital Equivalents.
Description: Hospital equivalents (HE) were defined to include the following events:
  1. Heart failure-related hospital admissions for 24 hours or longer
  2. Heart failure-related emergency department visits and necessitates invasive treatment (e.g. IV diuretic administration).
  3. Heart failure-related urgent visits and necessitates invasive treatment (e.g. IV diuretic administration).
Time Frame: 6 Months post-implant
Population: All randomized subjects
Measure: Mean (95% Confidence Interval); unit: Events
Arm/Group | Treatment | Control
Number analyzed (Participants) | 134 | 140
Events | 0.63 [0.51 to 0.78] | 0.81 [0.67 to 0.97]

4. Secondary Outcome: Health Care Utilization
Description: Characterize total health care utilization, the total number of all-cause hospitalization, emergency department, and urgent care visits.
Time Frame: 6 Months post-implant
Population: All randomized subjects
Measure: Number; unit: Total number of events
Arm/Group | Treatment | Control
Number analyzed (Participants) | 134 | 140
Total number of events | 218 | 255

5. Secondary Outcome: Days Hospitalization Free
Description: The number of days alive outside the hospital was calculated as the number of days of randomized follow-up minus the number of days hospitalized during the randomized follow-up period.
Time Frame: 6 Months post-implant
Population: All randomized subjects
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Treatment | Control
Number analyzed (Participants) | 134 | 140
Days | 170.8 [164.1 to 177.6] | 172.7 [166.6 to 178.9]

6. Secondary Outcome: Clinical Composite Response of Either "Worsened", "Improved", or "Unchanged"
Description: Worsened, Improved and Unchanged were defined as follows:
  Worsened: Patient died, hospitalized for worsening heart failure, worsened NYHA Class Improved: Patient improved in NYHA Class Unchanged: Patient was neither improved nor worsened.
Time Frame: 6 Months post-implant
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 134 | 140
Participants
  Improved | 56 | 48
  Worsend | 50 | 66
  Unchanged | 28 | 26

7. Secondary Outcome: Quality of Life Measured by the Minnesota Living With Heart Failure Questionnaire
Description: Quality of life was measured by the Minnesota Living with Heart Failure (MLHF), a questionnaire with 21 questions and scored on a scale from 0 (good quality of life) to 105 (low quality of life).
  Change in quality of life is defined as change from baseline to month 6. A participant must have completed a quality of life survey at the baseline visit and month 6 visit to be included in the analysis.
Time Frame: 6 Months post-implant
Population: All randomized subjects completing a quality of life survey at the baseline visit and month 6 visit
Measure: Mean (Full Range); unit: Index score
Arm/Group | Treatment | Control
Number analyzed (Participants) | 117 | 127
Index score | -12.5 [-69 to 42] | -8.5 [-73 to 89]

8. Secondary Outcome: New York Heart Association (NYHA) Class
Description: New York Heart Association (NYHA) Classifications were defined as follows:
  Class I - Patients with cardiac disease but without resulting limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or angina.
  Class II - Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or angina.
  Class III - Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or angina.
  Class IV - Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: 6 Months post-implant
Population: All randomized subjects with NYHA assessment completed at baseline and at 6 months were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 113 | 122
Participants
  NYHA I | 7 | 11
  NYHA II | 39 | 31
  NYHA III | 61 | 70
  NYHA IV | 6 | 10

9. Secondary Outcome: Distance Walked During a Six Minute Hall Walk
Description: Patients completed six minute hall walk at baseline and 6 months. Outcome is change in hall walk distance from baseline to 6 months.
Time Frame: 6 Months post-implant
Population: All randomized patients completing a hall walk at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Treatment | Control
Number analyzed (Participants) | 112 | 115
Meters | 6.2 (98.8) | -8.2 (114.2)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 13/134 | 11/140
Serious Adverse Events (participants affected / at risk) | 79/134 | 91/140
Other Adverse Events (participants affected / at risk) | 15/134 | 17/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=134) | Control (N=140)
Decompensation of heart failure (Cardiac disorders) | 35 (57) | 43 (68)
Volume overload (Cardiac disorders) | 6 (10) | 16 (26)
Volume depletion/dehydration (Cardiac disorders) | 6 (6) | 5 (6)
Angina pectoris (Cardiac disorders) | 8 (8) | 1 (1)
Cardiovascular procedure (Cardiac disorders) | 4 (4) | 5 (6)
Hypotension (Cardiac disorders) | 1 (1) | 4 (4)
Non-specific chest (Cardiac disorders) | 3 (4) | 4 (4)
Non sustained VT (Cardiac disorders) | 1 (1) | 3 (3)
Sustained VT (Cardiac disorders) | 1 (1) | 3 (3)
Acute MI/Cardiac Arrest (Cardiac disorders) | 3 (3) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Paroxysmal atrial flutter/fibrillation (Cardiac disorders) | 3 (4) | 1 (1)
Persistent atrial flutter/fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular fibrillation/flutter (Cardiac disorders) | 2 (2) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1) | 2 (2)
Renal insufficiencies/failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Electro Mechanical Dis-association (Cardiac disorders) | 0 (0) | 1 (1)
Hyponatremia (Endocrine disorders) | 0 (0) | 1 (1)
Hypokalemia (Endocrine disorders) | 0 (0) | 2 (2)
Elective Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Inhalant Poisoning from Cleaning Agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sudden Cardiac Death (Cardiac disorders) | 1 (1) | 1 (1)
Dyspnea/SOB (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Edema/weight gain (Cardiac disorders) | 1 (1) | 0 (0)
Lab value abnormalities (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Worsening COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (General disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Change in mental status (Psychiatric disorders) | 1 (2) | 0 (0)
Respiratory Failure/Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
MRSA Infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac Transplant (Cardiac disorders) | 1 (1) | 0 (0)
Peripheral Vascular Disease (Vascular disorders) | 1 (1) | 0 (0)
Allergic Reaction (General disorders) | 1 (1) | 0 (0)
Coronary Artery (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=134) | Control (N=140)
Sustained VT (Cardiac disorders) | 0 (0) | 2 (2)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0)
Decompensated Heart Failure (Cardiac disorders) | 5 (6) | 5 (5)
Angina (Cardiac disorders) | 2 (3) | 1 (1)
Volume depletion/dehydration (Cardiac disorders) | 2 (2) | 3 (3)
Volume overload (Cardiac disorders) | 4 (4) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No